CLINICAL TRIAL: NCT05986682
Title: Real-World Analysis of Belantamab Mafodotin Care Patterns in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00110976; 218855 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory; Ophthalmology; Keratopathy; Distress; National Comprehensive Cancer Network (NCCN) Distress Thermometer; Retrospective; Patient Reported Outcomes; Belantamab Mafodotin; Blenrep
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Blenrep — Belantamab Mafodotin - blmf (BLENREP) given for the treatment of relapsed and/or refractory multiple myeloma.

SUMMARY:
The purpose of this study is to describe the real-world use of Belantamab Mafodotin - blmf (BLENREP) and associated patterns of care, including dosing and dose modification, eye care specialist visits, associated healthcare utilization, and clinical outcomes in patients with relapsed and/or refractory multiple myeloma (RRMM) seen in the Duke Cancer Institute (DCI) clinics.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age as of start of treatment with BLENREP
* Patients with a corresponding diagnosis code consistent with multiple myeloma seen at Duke.
* Patients with a record of starting treatment with BLENREP for RRMM between August 5, 2020 and November 22, 2022.
* Patients having healthcare encounters at Duke Cancer Institute (DCI) for at least 1-month after start of Blenrep treatment.

Exclusion Criteria:

* Patients who were included in any clinical trial for BLENREP including expanded access clinical trials
* Age > 89 years of age as of start of index therapy

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will analyze clinical data from adult patients with relapsed and/or refractory multiple myeloma who were treated with Belantamab Mafodotin - blmf (BLENREP) in the DCI Oncology outpatient clinics between August 5, 2020 and November 7, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W LeBlanc, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel MN, Locke SC, Falvey C, Troy JD, Herring KW, Bolgioni-Smith A, Elcock C, Iadeluca L, Costa Chase C, Gasparetto C, Newman MS, LeBlanc TW. Treatment Patterns, Efficacy, and Tolerability of Belantamab Mafodotin in Patients With Relapsed and/or Refractory Multiple Myeloma: A Real-World Analysis. Clin Lymphoma Myeloma Leuk. 2025 Aug;25(8):e570-e579.e4. doi: 10.1016/j.clml.2025.04.008. Epub 2025 Apr 15. PMID 40348718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-site, retrospective, observational study examining longitudinal care patterns for belantamab mafodotin among relapsed and/or refractory multiple myeloma (RRMM) patients seen at Duke Cancer Institute (DCI).
Pre-assignment Details: 57 Duke patients were identified with RRMM who began treatment with Blenrep between Aug 5, 2020 and Nov 22, 2022. 25 patients were excluded (9 concurrently receiving other therapies, 8 being followed by a local oncologist or without Blenrep Risk Evaluation and Mitigation Strategies [REMS] documentation, 5 with <1 mo. of follow-up, and 3 receiving Blenrep as part of an expanded access pathway). Of the 32 remaining patients, 30 patients were randomly selected for chart abstraction.
Groups:
- Multiple Myeloma/Blenrep Participants: Participants with relapsed and/or refractory multiple myeloma who were treated with Belantamab Mafodotin - blmf (BLENREP) in the DCI Oncology outpatient clinics between August 5, 2020 and November 7, 2023.
Period: Overall Study
Arm/Group | Multiple Myeloma/Blenrep Participants
Started | 30
Completed (Completed is defined as having contributed data during the study period.) | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] — Age at Treatment Initiation (Baseline)
  years | 68 [45 to 87]
Age, Continuous [Median (Full Range); unit: years] — Age at Multiple Myeloma Diagnosis
  years | 61 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 14
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Current Payer type [Count of Participants; unit: Participants]
  Medicare + Commercial | 19
  Medicare + Military | 3
  Medicare + Medicaid | 1
  Commercial Alone | 6
  Medicaid Alone | 1
Diagnosis Location [Count of Participants; unit: Participants]
  At Duke | 15
  External Location | 15
Multiple Myeloma (MM) Diagnostic Characteristics [Count of Participants; unit: Participants] — Participants may have more than one diagnostic characteristic of MM.
  Participants
    >= 10% Bone Marrow Plasma Cells | 29
    Plasmacytoma (Total) | 9
    Bone Plasmacytoma | 8
    Extramedullary Plasmacytoma | 1
    >60% Bone Marrow plasma cells | 17
    ≥ 100 serum free light chain (FLC) ratio | 14
    >1 focal lesion on MRI | 5
    Hypercalcemia | 6
    Renal Insufficiency | 5
    Anemia | 17
    ≥ 1 Bone lesion (X-ray, CT, PET) | 21
MM Subtype - Immunoglobulin (Ig) [Count of Participants; unit: Participants] — Subtype of MM by Immunoglobulin - as determined at Diagnosis
  Participants
    IgG | 16
    IgA | 9
    IgD | 0
    IgE | 0
    IgM | 0
    Light Chain Only | 0
    Non-secretory | 5
MM Subtype - Involved Serum Free Light Chain [Count of Participants; unit: Participants] — Subtype of MM by involved serum free light chain - as determined at Diagnosis
  Participants
    Kappa | 18
    Lambda | 12
R-ISS Score [Count of Participants; unit: Participants] — The Revised International Staging System (R-ISS) is a prognostic staging system used to stratify patients with MM based on genetic risk as assessed by fluorescence in-situ hybridization (FISH) and routinely used lab values. The R-ISS system consists of stage I: serum beta2-microglobulin < 3.5 milligram per liter (mg/L), albumin >= 3.5 gram per deciliter (g/dL), standard-risk chromosomal abnormalities (CA) by FISH and normal lactate dehydrogenase level (LDH); stage II: neither R-ISS stage I nor stage III; and stage III: beta2-microglobulin >= 5.5mg/L and either high-risk CA by FISH or high LDH.
  Participants
    R-ISS I | 2
    R-ISS II | 5
    Unknown | 23
High Risk Abnormalities at Diagnosis [Count of Participants; unit: Participants] — High-Risk abnormalities identified by cytogenetic testing at diagnosis. International Myeloma Working Group (IMWG)- defined High Risk is the percentage of patients who had any of the following high risk traits: t(4;14), t(14;16), del(17p).
  Participants
    t(4;14) | 1
    t(14;16) | 2
    del(17p)/monosomy 17 | 4
    1q21 gain/amplification | 12
    t(14;20) | 1
    High Risk by IMWG | 7
Standard-Risk Abnormalities at Diagnosis [Count of Participants; unit: Participants] — Standard-Risk abnormalities identified by cytogenetic testing at diagnosis
  Participants
    t(6;14) | 0
    t(11;14) | 3
    MYC translocation | 3
    TP53 mutation | 0
    trisomies/tetrasomies | 12
    Complex karyotype (when done) or karyotypic del(13) | 14
Median Number of Lines of Therapy prior to Baseline [Median (Full Range); unit: Lines of therapy] | 4 [2 to 7]
Number of Prior Lines of Therapy - categorical [Count of Participants; unit: Participants]
  < 4 Lines of Therapy | 10
  ≥ 4 Lines of Therapy | 30
Types of Prior Therapy [Count of Participants; unit: Participants]
  Immunomodulatory Agents | 30
  Proteasome Inhibitors | 30
  Monoclonal Antibodies | 29
  Conventional Chemotherapy | 20
  Novel Agents | 13
  Stem Cell Transplant | 19
  Clinical Trials | 6
  Other | 2
Type of Refractory MM [Count of Participants; unit: Participants] — Represents the number of lines patients were refractory to - Double (2 lines), Triple (3), Quad (4) or Penta (5)
  Participants
    Double | 4
    Triple | 12
    Quad | 1
    Penta | 13
History of Prior Malignancy [Count of Participants; unit: Participants]
  Bladder | 1
  Brain and Spinal Cord | 1
  Breast | 1
  Kidney | 1
  Prostate | 1
  Skin Melanoma | 1
  Uterine | 1
  Smoldering MM | 5
  monoclonalgammopathy of unknown significance | 2
Baseline ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status as graded by clinician using the following Grades: 0: Fully active, able to carry on all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory, able to carry out work of light nature. 2: Ambulatory, capable of self-care, unable to carry out work activities. Up and about more than 50% waking hours. 3: Capable of limited self-care, confined to bed/chair more than 50% waking hours. 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed/chair. 5: Dead.
  Participants
    1 | 11
    2 | 3
    3 | 1
    Unknown | 15
Baseline Renal Impairment [Count of Participants; unit: Participants] — Baseline Renal Impairment - Estimated Glomerular Filtration Rate (eGFR)
  Participants
    Normal | 2
    Mild | 16
    Moderate | 10
    Severe | 2
Baseline Renal Impairment (as measured by Serum Creatinine levels) [Count of Participants; unit: Participants] — Serum Creatinine levels are used here as a measure of renal function. For this study, renal insufficiency is defined as a baseline serum creatinine level of >= 2.0 mg/dL.
  Participants
    Serum Creatinine ≥ 2.0 mg/dL | 3
    Serum Creatinine < 2.0 mg/dL | 27

OUTCOME MEASURES:

1. Primary Outcome: Treatment Characteristics: Duration of Treatment With BLENREP
Description: Duration of Treatment Duration calculated from first Blenrep dose to either treatment discontinuation (for subjects who discontinued treatment prior to study end date) or last dose (for subjects who were continuing treatment as of study end date). Descriptive statistics consisting of the median (with interquartile range) was used to summarize duration across participants.
Time Frame: Between baseline and earliest of end of BLENREP treatment, death, lost to contact or end of study timeframe, up to 40 months.
Population: All patients were analyzed.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Months | 9.3 [0.7 to 21.6]

2. Primary Outcome: Treatment Characteristics: Discontinuation of BLENREP Treatment
Description: Number of participants who discontinued treatment with BLENREP by reason.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Discontinuations for any reason | 26
  Discontinuation for Disease Progression | 22
  Discontinuation for Corneal or other ocular toxicity | 4
  Discontinuation for Physician/Patient choice | 3
  Discontinuation for other reason | 3

3. Primary Outcome: Treatment Characteristics: Dosing Patterns - Number of Cycles of Treatment With BLENREP Therapy
Description: Treatment characteristics: Dosing patterns - Number of cycles of treatment with BLENREP therapy - From Treatment initiation to treatment discontinuation or last dose during study period.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Cycles
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Cycles
  Total # of cycles | 6.5 [2 to 13]
  # of cycles at 2.5 mg/kg^2 | 2 [1 to 11]
  # of cycles at 1.9 mg/kg^2 | 3 [1 to 11]

4. Primary Outcome: Treatment Characteristics: Dosing Patterns - Delays in Treatment With BLENREP Therapy
Description: Number of participants for whom BLENREP dosing was delayed during treatment as categorized by reason.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Delay for any reason | 27
  Delay for Corneal AE | 27
  Delay for Other Ocular Toxicity | 2
  Delay for Hematologic Toxicity | 3
  Delay for Physician/Patient Choice | 2
  Delay for any other reason | 10

5. Primary Outcome: Treatment Characteristics: Dosing Patterns - Dose Reductions During Treatment With BLENREP Therapy
Description: Number of participants for whom BLENREP dosing was dose reduced during treatment as categorized by reason.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Total # of Participants with Dose Reductions for Any Reason | 19
  Dose Reduction for Corneal Adverse Event | 13
  Dose Reduction for Hematologic Toxicity | 6
  Dose Reduction for Other Reason | 1

6. Primary Outcome: Clinical Outcomes: Best Overall Response
Description: Response categorized using modified IMWG 2016 criteria. Urine testing was not routinely done; only serum M-protein levels were used when determining response. Complete Response(CR)= negative immunofixation on the serum + absence of any soft tissue plasmacytomas + <5% plasma cells in bone marrow aspirates. Very Good Partial Response(VGPR) = serum detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein. Partial Response(PR) = ≥50% reduction of serum M-protein. If the serum is unmeasurable, a > 50% decrease in the difference between involved and uninvolved FLC levels is required. Stable Disease (SD) = not meeting criteria for CR, VGPR, PR, or progressive disease. Progressive Disease (PD) = >25% increase from lowest response value in serum M-protein (the absolute increase must be >0.5 g/dL), or definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  CR | 0
  VGPR | 11
  PR | 9
  SD | 9
  PD | 1

7. Primary Outcome: Clinical Outcomes: Time To Response
Description: The time from the start of BLENREP treatment to the date of first occurrence of response (partial response or better).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Months | 1.4 [0.7 to 3.8]

8. Primary Outcome: Clinical Outcomes: Time To Best Response
Description: The time from the start of BLENREP treatment to the date of the best response achieved (partial response or better).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Months | 1.5 [0.7 to 9.9]

9. Primary Outcome: Clinical Outcomes: Duration of Response
Description: The time from the first date of PR or better to the earliest of documented disease progression, end of BLENREP treatment, death, lost to followup or end of study timeframe.
Time Frame: as for outcome 1
Population: Analyzed only for the 20 patients who achieved PR or better
Measure: Median (Full Range); unit: Months
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 20
Months | 9.8 [1.1 to 20.2]

10. Primary Outcome: Clinical Outcomes: Progression-Free Survival (PFS)
Description: The time from the start of BLENREP treatment until the earliest of documented disease progression (according to IMWG response criteria or clinician assessment), end of BLENREP treatment, death, lost to followup or end of study timeframe.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Months | 8.4 [6.6 to 12.7]

11. Primary Outcome: Clinical Outcomes: Overall Survival (OS)
Description: Summary report of patient status at the end of the study period. Duration of survival was calculated, however, median survival time for OS has not yet been reached, and therefore is not reported here.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Alive | 19
  Deceased | 10
  Unknown/Lost to Follow Up | 1

12. Secondary Outcome: Ophthalmology: Presence of Ocular Toxicity
Description: Number of participants with specific ocular events of interest during treatment with BLENREP
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Number of Participants with a Corneal Event | 28
  Number of Participants with a change to Best-Corrected Visual Acuity | 27

13. Secondary Outcome: Ophthalmology: Number of Ocular Toxicity Events Per Participant
Description: Number of Ocular Toxicity Events (Corneal Event or Best-Corrected Visual Acuity Change) per patient, summarized by median (min, max).
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Events
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Events
  Number of Corneal Events | 10.5 [2 to 25]
  Number of changes to Best-Corrected Visual Acuity | 7 [1 to 25]

14. Secondary Outcome: Ophthalmology: Treatments for Ocular Toxicity
Description: Number of participants receiving treatment for ocular toxicity during BLENREP therapy, as categorized by type of treatment.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Received any Treatment for Ocular Toxicity | 30
  Encouraged Adherence to Eye Drop Regimen | 15
  Increased Eye Drops | 10
  Received a new prescription - Eye drops/ointment | 11
  Other | 1

15. Secondary Outcome: Magnitude of Distress Using National Comprehensive Cancer Network Distress Thermometer (NCCN DT)
Description: Distress is measured on a scale of 0-10 on the National Comprehensive Cancer Network Distress Thermometer (NCCN DT). A score of 0 represents no distress, and a score of 10 represents worst possible distress. Actionable distress is defined as a NCCN DT score of 4 or higher, and is aligned with the medical practice guidelines for management of distress in cancer patients.The median (min, max) distress score across patients is reported.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: DT Score
Units Other Than Participants: Scores
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Scores) | 194
DT Score | 1.33 [0.00 to 7.56]

16. Secondary Outcome: Sources of Distress Using NCCN DT: Frequency of Reported Problems
Description: Sources of distress will be assessed using the NCCN DT Problem List by examining the percentage of visits where types of problems are reported. There are five categories of distress from which patients can report problems (practical, family, emotional, physical and other problems). The categories of problems are reported as a number and % of the total number of visits where problem lists are reported.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Visits) | 209
Visits
  Practical Problems | 27
  Family Problems | 17
  Emotional Problems | 46
  Physical Problems | 107
  Other Problems | 23

17. Secondary Outcome: Sources of Distress Using NCCN DT: Top 5 Most Frequently Reported Problems
Description: Sources of distress will be assessed using the NCCN DT Problem List by examining the percentage of visits where types of problems are reported. The problem list includes 39 possible problems from which patients can choose. The problems are reported as a number and % of the total number of visits where problem lists are reported.
Time Frame: as for outcome 1
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Visits) | 209
Visits
  Fatigue | 69
  Pain | 63
  Tingling in Hands/Feet | 40
  Worry | 33
  Getting Around | 31

18. Secondary Outcome: Healthcare Resource Utilization (HCRU)
Description: To the extent that they are available, HCRU [i.e., radiation therapy, transfusions (red blood cells or platelets), inpatient admissions, treatment-related outpatient visits, emergency department visits, palliative care outpatient visits] that occurred during BLENREP treatment will be summarized by the percentage and frequency distribution of patients with any occurrence of the respective outcome.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Participants
  Received Radiation Therapy | 3
  Transfusions | 7
  Inpatient Admissions | 10
  Treatment-Related Outpatient Visits | 20
  Emergency Department Visits | 11
  Palliative Care Outpatient Visit | 10

19. Post Hoc Outcome: Ophthalmology: Number of Ocular Symptoms Reported
Description: Study procedures included recording ocular symptoms reported by patients documented in the clinic notes. These were categorized into blurry vision, dry eyes, photophobia and other symptoms (including foreign-body sensation, "grittiness", "itch/scratchiness", irritation, and tearing). This Data table reports the total number of Ocular Symptoms reported by patients, along with counts and percentage by type of symptom.
Time Frame: as for outcome 1
Population: The 30 patients in the study reported specific symptoms a total of 192 times at clinic visits. The analysis population is the 192 symptoms reported.
Measure: Count of Units; unit: Ocular Symptoms
Units Other Than Participants: Ocular Symptoms
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Ocular Symptoms) | 192
Ocular Symptoms
  Number of Ocular Symptoms reported | 192
  Blurry Vision | 102
  Dry Eyes | 32
  Photophobia | 26
  Other | 32

20. Post Hoc Outcome: Ophthalmology: Grade of Ocular Toxicities (Corneal Events)
Description: Ocular toxicity as measured by corneal events per the Keratopathy Visual Acuity scale, and graded using belantamab mafodotin REMS [Risk Evaluation and Mitigation Strategies] guidelines. Corneal examination changes from baseline are categorized as normal or grade 1, 2, 3, or 4 and are based on the worst overall finding. Normal: Cornea clear/No change from baseline. Grade 1: Mild superficial keratopathy with or without symptoms. Grade 2: Moderate superficial keratopathy. Grade 3: Severe superficial keratopathy. Moderate/Severe keratopathy could be with or without patchy microcyst-like deposits, sub-epithelial haze (peripheral), or a new peripheral stromal opacity. Grade 4: Corneal epithelial defect (such as corneal ulcer). The Data table reports the total number of corneal events experienced, along with counts and percentage by grade of event.
Time Frame: as for outcome 1
Population: The 30 patients in the study experienced ocular toxicity (corneal events) a total of 323 times as reported during clinic visits. The analysis population is the 323 events reported.
Measure: Count of Units; unit: Corneal Events
Units Other Than Participants: Corneal Events
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Corneal Events) | 323
Corneal Events
  Total Number of Corneal Events | 323
  Grade 1 | 158
  Grade 2 | 158
  Grade 3 | 4
  Grade 4 | 3

21. Post Hoc Outcome: Ophthalmology: Time to Resolution of Clinically Meaningful Ocular Toxicities - Corneal Events
Description: Clinically Meaningful Event is defined as an event that is grade >= 2 for which BLENREP administration is halted until the event resolves to grade <= 1. Time to resolution is calculated for events that resolved. Unresolved events are those that had not returned to grade <=1 at last contact due to either end of study or lost to ophthalmologic follow-up. There were 64 resolved events for Corneal Events that were analyzed
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Units Other Than Participants: Resolved Events
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Resolved Events) | 64
Weeks | 6 [2 to 22]

22. Post Hoc Outcome: Ophthalmology: Grade of Ocular Toxicities [Changes to Best-Corrected Visual Acuity (BCVA)]
Description: Ocular toxicity as measured by changes to BVCA as measured per the Keratopathy Visual Acuity scale, and graded using belantamab mafodotin REMS [Risk Evaluation and Mitigation Strategies] guidelines. BVCA changes from baseline are categorized as normal or grade 1, 2, 3, or 4 and are based on the worst overall finding. Normal: No decline from baseline on Snellen Visual Acuity. Grade 1: Decline from baseline of 1 line on Snellen Visual Acuity. Grade 2: Decline from baseline of 2 or 3 lines on Snellen Visual Acuity, and not worse than 20/200. Grade 3: Decline from baseline of more than 3 lines on Snellen Visual Acuity, and not worse than 20/200. Grade 4: Snellen Visual Acuity worse than 20/200. The Data table reports the total number of BVCA changes experienced, along with counts and percentage by grade of change.
Time Frame: as for outcome 1
Population: The 30 patients in the study experienced ocular toxicity (changes to BVCA) a total of 244 times as reported during clinic visits. The analysis population is the 244 BVCA changes reported.
Measure: Count of Units; unit: BVCA Changes
Units Other Than Participants: BVCA Changes
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (BVCA Changes) | 244
BVCA Changes
  Total Number of Changes to BVCA | 244
  Grade 1 | 125
  Grade 2 | 111
  Grade 3 | 8
  Grade 4 | 0

23. Post Hoc Outcome: Ophthalmology: Time to Resolution of Clinically Meaningful Ocular Toxicities - Best Corrected Visual Acuity
Description: Clinically Meaningful Event is defined as an event that is grade >= 2 for which BLENREP administration is halted until the event resolves to grade <= 1. Time to resolution is calculated for events that resolved. Unresolved events are those that had not returned to grade <=1 at last contact due to either end of study or lost to ophthalmologic follow-up. There were 44 Resolved events for changes in Best Corrected Visual Acuity that were analyzed.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: Weeks
Units Other Than Participants: Resolved Events
Arm/Group | Multiple Myeloma/Blenrep Participants
Number analyzed (Participants) | 30
Number analyzed (Resolved Events) | 44
Weeks | 6 [3 to 53]

24. Post Hoc Outcome: Hospice Care Given Prior to Death
Description: The number and percentage of patients who were in Hospice Care prior to death. Analyzed for the 10 patients who died as of last follow-up Dec. 1st 2023.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Multiple Myeloma/Blenrep Participants Who Died: Participants with relapsed and/or refractory multiple myeloma who were treated with Belantamab Mafodotin - blmf (BLENREP) in the DCI Oncology outpatient clinics between August 5, 2020 and November 7, 2023; and who died prior to December 1, 2023.
Arm/Group | Multiple Myeloma/Blenrep Participants Who Died
Number analyzed (Participants) | 10
Participants
  Yes | 4
  No | 5
  Unknown | 1

ADVERSE EVENTS:
Time Frame: Between baseline and earliest death, lost to contact or end of study timeframe, up to 40 months.
Description: Ocular AEs were collected per participant, not per eye. Hematologic toxicity was collected if it was a reason for change to treatment. No other AEs were collected. Ocular toxicity was collected systematically through optometrist visits; measured per the Keratopathy Visual Acuity scale, using belantamab mafodotin REMS guidelines. Ocular symptoms were reported ad hoc by patients at individual clinic visits, as a non-systematic assessment. Serious AEs were not monitored/assessed.
Arm/Group | Multiple Myeloma/Blenrep Participants
All-Cause Mortality (participants affected / at risk) | 10/30
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 29/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Myeloma/Blenrep Participants (N=30)
Keratopathy (Eye disorders) | 28 (320) — Ocular adverse events were collected per participant, not per eye.
Corneal epithelium defect (Eye disorders) | 3 (3) — Ocular adverse events were collected per participant, not per eye.
Visual acuity reduced (Eye disorders) | 27 (244) — Ocular adverse events were collected per participant, not per eye.
Blurred vision (Eye disorders) | 24 (102) — Ocular adverse events were collected per participant, not per eye.
Dry eye (Eye disorders) | 9 (32) — Ocular adverse events were collected per participant, not per eye.
Photophobia (Eye disorders) | 9 (26) — Ocular adverse events were collected per participant, not per eye.
Foreign body sensation in the eye (Eye disorders) | 4 (6) — Ocular adverse events were collected per participant, not per eye.
Eye pruritus (Eye disorders) | 2 (10) — Ocular adverse events were collected per participant, not per eye.
Eye pain (Eye disorders) | 3 (5) — Ocular adverse events were collected per participant, not per eye.
Eye irritation (Eye disorders) | 7 (9) — Ocular adverse events were collected per participant, not per eye.
Lacrimation increased (Eye disorders) | 1 (1) — Ocular adverse events were collected per participant, not per eye.
Ocular discomfort (Eye disorders) | 1 (1) — Ocular adverse events were collected per participant, not per eye.
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Abnormal LFT (liver function test) (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05986682/Prot_SAP_000.pdf